CLINICAL TRIAL: NCT03543995
Title: The Relationship Between Nocturnal Enuresis And Spina Bifida Occulta: A Prospective Controlled Trial
Brief Title: The Relationship Between Nocturnal Enuresis And Spina Bifida Occulta
Status: Completed | Type: Observational
Sponsor: Ankara Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Muhammet Fatih Kilinc, Principal Investigator, Ankara Training and Research Hospital
Other Study IDs: 5520
Record Dates: First submitted 2018-05-22; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Enuresis, Nocturnal; Spina Bifida
Keywords: lower urinary tract symptoms; nocturnal enuresis; spina bifida occulta; treatment response
MeSH Terms: conditions — Nocturnal Enuresis; Spinal Dysraphism; Lower Urinary Tract Symptoms; Spina Bifida Occulta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Enuresis nocturna: Patients aged 6 to 15 years with at least one night-time wetting weekly
- Normal population: Patients who were admitted to the urology clinic with a complaint of abdominal or lateral pain, who had no NE and had a direct abdominal x-ray examination

SUMMARY:
It is claimed that SBO may be responsible for bladder dysfunction in patients without known neurological disease. Subsequently, it was reported that the frequency of SBO in NE cases was higher than normal children. However, in controlled trials, SBO frequency was not different in NE patients compared to the normal population. Conversely, the incidence of dysfunctional bladder in the presence of SBO in NE patients was found to be higher and the response to treatment was worse than in non-SBO patients.

The present study aimed to determine whether the frequency of SBO in patients with NE was higher than in healthy subjects, the effect of SBO on the severity of LUTS and whether treatment response of primary NE patients changed in the presence of SBO.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 6 to 15 years
* at least one night-time wetting weekly

Exclusion Criteria:

* neurological disease,
* diabetes mellitus or insipidus,
* spinal surgery history, spina bifida skin findings,
* chronic renal insufficiency
* and secondary enuresis

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients aged 6 to 15 years who were admitted to an urology outpatient clinics with at least one night-time wetting weekly, were included in this prospective study.
  The control group consisted of patients who were admitted to the urology outpatient clinic with a complaint of abdominal or lateral pain, who had no NE and had a direct abdominal x-ray examination. The patients who were selected as the control group had night wetness questioned and the dysfunctional voiding symptom score (DVSS) form was completed. Those who had night wetting, neurological disease or diabetes mellitus were not included in the control group.
Sampling Method: Non-Probability Sample
Enrollment: 330 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-15 (Actual)

PRIMARY OUTCOMES:
Dry bed days | 3 months
  Patients were called for check-up one and three months later. When waking in the morning they were given a form to mark as dry or wet, and dry bed days were examined at check-up.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Kurt O, Yazici CM, Paketci C. Nocturnal enuresis with spina bifida occulta: Does it interfere behavioral management success? Int Urol Nephrol. 2015 Sep;47(9):1485-91. doi: 10.1007/s11255-015-1047-4. Epub 2015 Jul 7. PMID 26149636
- [Result] Cakiroglu B, Tas T, Eyyupoglu SE, Hazar AI, Can Balci MB, Nas Y, Yilmazer F, Aksoy SH. The adverse influence of spina bifida occulta on the medical treatment outcome of primary monosymptomatic nocturnal enuresis. Arch Ital Urol Androl. 2014 Dec 30;86(4):270-3. doi: 10.4081/aiua.2014.4.270. PMID 25641449
- [Result] Miyazato M, Sugaya K, Nishijima S, Owan T, Ogawa Y. Location of spina bifida occulta and ultrasonographic bladder abnormalities predict the outcome of treatment for primary nocturnal enuresis in children. Int J Urol. 2007 Jan;14(1):33-8. doi: 10.1111/j.1442-2042.2006.01666.x. PMID 17199857